CLINICAL TRIAL: NCT07147283
Title: Study Protocol, Increasing Awareness and Early Detection in Students at Risk of Gynaecological Cancer: Feasibility of an Online Educational and Behaviour Change Intervention
Brief Title: Protocol: Feasibility of an Online Intervention to Increase Awareness of Gynaecological Cancer in UK Students
Acronym: GoCheck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leeds Beckett University (Other)
Responsible Party: Principal Investigator, Trish Holch, Professor of Applied Health Psychology, Leeds Beckett University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HOLCH_EVE_APPEAL; EVE/0032 (Other Grant/Funding Number: The Eve Appeal)
Record Dates: First submitted 2025-08-13; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Intervention
Keywords: Behaviour change; Theory of planned behaviour; Gynaecological Cancer; Volitional help sheet; Educational film

STUDY DESIGN:
Intervention Model Description: Design This is a randomised mixed methods feasibility study with repeated measures and adheres to the Medical Research Council (MRC) guidance on the development, implementation, and evaluation of complex health care interventions. Young women (or transexual or non- binary individuals with female anatomy) at UK universities will be randomised with 1:1 allocation to either an intervention (an online gynaecological cancer awareness film and volitional help sheet implementation behaviour change intervention) or the control condition via the randomisation facility in Qualtrics™.
  Cancer awareness and plans for self-monitoring will be assessed at baseline, 4 weeks, 3 months and 6 months, along with assessment of the theory of planned behaviour domains (supplementary information 2). Feasibility of the intervention will be assessed by recruitment and retention rates and qualitative interviews.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No cancer awareness film and help sheet (No Intervention): Participants assigned to the control condition will have no exposure to cancer education over and above what is available generally and be assessed on their previously accrued cancer information. They will take part in the study and complete the questionnaires at baseline, 4 weeks, 3 months and 6 months.
- Intervention: cancer awareness film and help sheet (Experimental): The intervention consists of a bespoke online gynaecological cancer awareness educational film and a volitional help sheet to plan future gynaecological help seeking and monitoring based on implementation intention principles. The intervention will be delivered online using Qualtrics™.
  Interventions: Behavioral: Educational film and volitional help sheet

INTERVENTIONS:
Behavioral: Educational film and volitional help sheet — The intervention consists of a bespoke online gynaecological cancer awareness educational film and a volitional help sheet to plan future gynaecological help seeking and monitoring based on implementation intention principles [24]. The intervention will be delivered online using Qualtrics™.
  Arms: Intervention: cancer awareness film and help sheet

SUMMARY:
In the UK more than 2500 young people are diagnosed with cancer each year, including gynaecological cancers) and almost a third will be diagnosed within accident and emergency departments. Early diagnosis is essential to improve cancer outcomes. However, despite awareness of warning signs, most young people would delay or avoid seeking help altogether. The key to lifelong monitoring and early detection of cancer is early exposure to cancer information at a formative age. University is seen as a key life transition phase which will enable students to establish positive health behaviours.

We have developed an online intervention to change behaviour for university students to support the early detection and intention to seek help for symptoms of gynaecological cancer. The intervention consists of a gynaecological cancer awareness educational film and a help sheet to plan future help seeking. The aim of this study is to find out if the intervention is acceptable for participants and practicable to run.

Methods We aim to recruit 86 participants who are women (or those at risk of gynaecological cancer e.g., have ovaries, a uterus, cervix) over 18 at UK universities who can understand English. The educational film provides information about the signs and symptoms of the five different forms of gynaecological cancer and will be delivered online to participants. The help sheet encourages participants to self-monitor for gynaecological symptoms and then identify cues to help-seeking/action. Cancer awareness and willingness to seek help for symptoms will be assessed by questionnaires four times at the beginning, and at 4 weeks, 3 months and 6 months). Interviews will be carried out with participants to understand how acceptable the intervention is.

Results Acceptability will be measured by looking at how many people have been recruited and how many have dropped out of the study, how long they have taken to watch the film and to complete the help sheet. Interviews will be analysed by theme.

Conclusion We hope that the findings from this study will provide evidence of how the intervention can increase cancer awareness and likelihood of help seeking for cancer symptoms. The long-term goal is to use these findings to use this intervention in other universities in the UK.

DETAILED DESCRIPTION:
Background In the UK more than 2500 Teenage and Young Adult (TYA) are diagnosed with cancer each year, the majority being melanomas or carcinomas (including gynaecological cancers). Alarmingly, almost a third (29%) of TYA cancers are diagnosed within accident and emergency departments. Early diagnosis is key to improved cancer outcomes. However, although a sample of university students, could identify the common cancer warning signs, (e.g. lumps, bleeding) they could not identify those less common including; constipation, frequency in urination and bloating. Further, despite awareness of warning signs, most young people would delay or avoid seeking help altogether. The key to lifelong monitoring and early detection of cancer is early exposure to cancer information and body awareness at a formative age. University is seen as a key life transition phase which will enable students to establish positive health behaviours.

We have developed an online behaviour change intervention for university students to support the early detection and intention to seek help for symptoms of gynaecological cancer. The intervention consists of a bespoke online gynaecological cancer awareness educational film and a volitional help sheet to plan future gynaecological help seeking. Aim: To establish the feasibility and acceptability of the intervention and to understand the barriers and enablers to uptake and how to improve the intervention to develop a definitive study for launch in UK Universities.

Methods A longitudinal 1:1 randomised mixed methods feasibility study design will be employed. Eligible participants are women (or those at risk of gynaecological cancer e.g., have ovaries, a uterus, cervix) over 18 at UK universities who can understand English. We aim to recruit N=86 participants online from UK Universities. The educational film provides information about the signs and symptoms of the five different forms of gynaecological cancer and will be delivered online to participants via Qualtrics™. The volitional help sheet encourages participants to self-monitor for gynaecological symptoms and then use a standard implementation intention exercise to identify cues to help-seeking/action. Cancer awareness will be assessed by the Young Person's Cancer Awareness Measure (YPCAM) at baseline, 4 weeks, 3 months and 6 months, along with assessment of the Theory of Planned Behaviour (TPB) domains. Semi-structured interviews with a subsection of the intervention group will explore the barriers and enablers to uptake.

Results Feasibility will be measured by assessing the proportion of recruitment and attrition rates per time point, study completion and adherence to the educational film and volitional help sheet. Mean score changes (intervention vs control) will be examined over the four timepoints adjusting for a single covariate (baseline scores). Interview data will be analysed using the six stages of reflexive thematic analysis. Progression criteria to a main trial would be the successful recruitment of 80% of the target sample.

Conclusion We hope the findings from this study will provide empirical evidence on the potential of the intervention to enhance cancer awareness and help-seeking behaviours for symptoms of gynaecological cancer among TYA. The long-term goal is to harness the insight gained form this study to provide evidence-based data that support the broader integration of open cancer awareness initiatives within university settings.

ELIGIBILITY:
Inclusion Criteria:

* female students (or those at risk of gynaecological cancer e.g., have ovaries, a uterus, cervix).
* over 18 years of age
* attending UK universities
* resident in the UK
* able to understand written English.

Exclusion Criteria:

* non- female students and those who are not at risk of gynaecological cancer e.g. (don't have ovaries, a uterus, cervix)
* under 18 years of age
* non UK residents
* not able to understand written English

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
Young Person Cancer Awareness Measure | From enrolment to 6 months
  Young Person's Cancer Awareness Measure (YPCAM) (supplementary information 1) at Baseline, 4-weeks, 3, 6 months. This 10-item measure is based on the adult Cancer Awareness Measure (CAM). Validated in adults (aged 18), assessing knowledge of cancer types, incidence rates, warning signs/symptoms and risk factors, and explores help-seeking intervals, past experience, and potential help-seeking barriers. A further iteration of this instrument (the YPCAM for TYA ≥16) was developed by the Teenage Cancer Trust and Dr Martin McCabe University of Manchester and includes the addition of advocacy and decision-making questions and has been utilised in UK studies However, the YPCAM has not yet been formally validated in TYA and therefore this limits the reliability of the findings. Scores range from one to five with five showing greater cancer awareness and willingness to help seek.

SECONDARY OUTCOMES:
Theory of Planned Behaviour | From enrolment to the end of 6 months
  Theory of Planned Behaviour (TPB) (supplementary information 2) questionnaire at Baseline, 4-weeks, 3, 6 months. The TPB is the most widely used effective model in predicting intention, stating that intention is the precursor of behaviour. We have developed a questionnaire incorporating these factors based around a cervical cancer questionnaire used with young women in Ireland. This will explore participants attitudes, intentions, subjective norms, anticipated regret and perceived behavioural control in relation to cancer awareness and help-seeking. Scores on the TPB range from questionnaire range from 1-7 and lower scores within each of the domains translate to increased positive attitudes from themselves and friends and family; greater perceived behavioural control and behavioural intentions and greater anticipated regret.

CONTACTS AND LOCATIONS:
Overall Officials: Trish Holch, PhD, Principal Investigator — Leeds Beckett University
Locations (1):
- Leeds Beckett University, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared due to ethical reasons.